CLINICAL TRIAL: NCT02029924
Title: A Double-blinded, Randomised, Two -Period Crossover Euglycemic Clamp Trial Investigating the Pharmacokinetics, Glucodynamics and Safety of BioChaperone Insulin Lispro and Insulin Lispro (Humalog®) in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BC3-CT006
Record Dates: First submitted 2013-12-16; First posted 2014-01-08 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2014-09

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BioChaperone insulin lispro (Experimental): BioChaperone insulin lispro
  Interventions: Drug: BioChaperone insulin lispro
- Humalog® (Active Comparator): Humalog®
  Interventions: Drug: Humalog®

INTERVENTIONS:
Drug: BioChaperone insulin lispro — Single dose of 0.2 U/Kg body weight injected subcutaneously (under the skin)
  Arms: BioChaperone insulin lispro
Drug: Humalog® — Single dose of 0.2 /Kg body weight injected subcutaneously (under the skin)
  Arms: Humalog®

SUMMARY:
The addition of Biochaperone to insulin lispro may accelerate the onset and shorten the duration of action of insulin lispro due to a facilitation of the absorption of the insulin after subcutaneous injection.

The aim of the trial is to assess the efficacy and safety of BioChaperone insulin lispro in subjects with Type 1 diabetes under a dose of 0.2 U/Kg.

This trial is a single-center, randomised, double-blinded, two-treatment, two-period cross-over, 6-hour euglycaemic glucose clamp trial in subjects with Type 1 diabetes mellitus. Each subject will be randomly allocated to a single dose of BioChaperone insulin lispro 0.2 U/Kg and a single dose of Humalog® 0.2 U/Kg on 2 separate dosing visits.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 12 months.
* Treated with multiple daily insulin injections or insulin pump for at least 12 months.
* Body Mass Index (BMI): 18.0-28.0 Kg/m².

Exclusion Criteria:

* Type 2 diabetes mellitus.
* Receipt of any investigational product within 3 months prior to first dosing.
* Clinically significant abnormalities as judged by the investigator.
* Any systemic treatment with drugs known to interfere with glucose metabolism.
* History of alcoholism, or drug/chemical abuse as per Investigator's judgement.
* Use of tobacco or nicotine-contained product within 5 years prior to screening.
* Blood or plasma donation in the past month or more than 500 mL within 3 months prior to screening.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) | 30 minutes
  Area under the curve of the insulin lispro concentration - time curve from 0 to 30 minutes

SECONDARY OUTCOMES:
Pharmacokinetics: Early t0.5max(Lisp) | up to 6 hours post administration of study drug
  Time to first observed half maximum observed insulin lispro concentration
Glucodynamics: Area under the glucose infusion rate - time curve from t=0 to 6 hours | 6 hours
Glucodynamics: Early t0.5(GIRmax) | 6 hours
  Time to first observed half maximum glucose infusion rate
Glucodynamic: GIRmax (Maximum glucose infusion rate) | 6 hours
Pharmacokinetics: Area under the insulin lispro serum concentration. Time curve from t=0 to 6 hours | 6 hours
Pharmacokinetics: tmax(Lisp) - Time from t=0 hours to maximum observed insulin lispro concentration | 6 hours
Safety and Tolerability: adverse events, local tolerability, vital signs variation, ECG, laboratory safety parameters | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Neuss, Germany